CLINICAL TRIAL: NCT03919929
Title: Treating PCOS With Semaglutide vs Active Lifestyle Intervention
Acronym: TEAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0636; 1R01DK120612-01A1 (NIH)
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: PCOS; Adolescent Obesity; NAFLD
Keywords: Insulin Resistance
MeSH Terms: conditions — Pediatric Obesity; Non-alcoholic Fatty Liver Disease; Insulin Resistance | interventions — semaglutide; Diet, Reducing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diet Intervention (Active Comparator): Weight loss with dietary intervention
  Interventions: Other: Weight loss diet
- GLP-1 Intervention (Experimental): Participants will take a daily oral tablet of semaglutide for 4 months.
  Interventions: Drug: Semaglutide 3mg and 7mg [Rybelsus]

INTERVENTIONS:
Drug: Semaglutide 3mg and 7mg [Rybelsus] — Once daily oral tablet of semaglutide for 4 months
  Other Names: GLP-1 receptor agonist
  Arms: GLP-1 Intervention
Other: Weight loss diet — Prescribed weight loss diet to match weight loss in Drug arm
  Arms: Diet Intervention

SUMMARY:
Girls with obesity and polycystic ovarian syndrome will receive either glucagon like peptide-1 receptor agonist therapy or a dietary intervention for 12 weeks to decrease the metabolic syndrome, in particular to lower hepatic fat and improve insulin sensitivity.

DETAILED DESCRIPTION:
In obese girls with polycystic ovarian syndrome, testosterone and obesity combine to create unique pathology to increase metabolic disease including fatty liver and insulin resistance, which may be mediated by altered glucagon like peptide-1 activity. The investigators will treat girls with obesity and polycystic ovarian syndrome for 4 months with a glucagon like peptide-1 receptor agonist compared to dietary intervention to primarily lower hepatic fat and secondarily improve whole body and adipose insulin sensitivity. Mechanisms of hepatic metabolism, including rates of de novo lipogenesis and relative mitochondrial flux will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary- less than 2 hours of moderate (jogging, swimming etc) exercise a week.
2. BMI equal or greater than the 90th percentile for age and gender
3. PCOS per the most stringent NIH criteria adapted for adolescents (irregular menses >12 months post-menarche and clinical or biochemical hypertestosteronemia
4. Participants cannot be on hormonal contraception, so participants should remain abstinent or use reliable non-hormonal contraception (e.g. copper IUD) for the entire study period. For participants who receive semaglutide, they should avoid pregnancy for at least 2 months after stopping medication to avoid fetal exposure to the medication.

Exclusion Criteria:

1. Diagnosed with or have a family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2). Family history of medullary thyroid cancer or thyroid nodule palpated by endocrinologist at screening.
2. Use of medications known to affect insulin sensitivity: metformin (cannot have been used in the 3 months prior to screening), oral glucocorticoids within 10 days, atypical antipsychotics, immunosuppressant agents, HIV medications, hormonal contraception (cannot have been used in the 6 months prior to screening). Dermal patch or vaginal ring contraception methods.Weight loss medications or stimulants. Use of other products containing other GLP-1 agonists.
3. Currently pregnant or breastfeeding women. Development of pregnancy during the study period will necessitate withdrawal from the study.
4. Severe illness requiring hospitalization within 60 days.
5. Diabetes, defined as Hemoglobin A1C > 6.4%
6. BMI percentile less than the 90th percentile for age and sex. Weight >325 lbs. or <84 lbs.
7. Anemia, defined as Hemoglobin < 11 mg/dL
8. Diagnosed major psychiatric or developmental disorder limiting informed consent.
9. Implanted metal devices that are not compatible with MRI
10. Use of blood pressure medications.
11. Known liver disease other than NAFLD or AST or ALT >100 IU/L.
12. Personal history of pancreatitis
13. Known renal disease of any severity or an eGFR at screening of <45ml/min/1.73m2
14. History of severe GI disease (e.g. gastroparesis)
15. History of gallstones
16. Untreated thyroid disease
17. History of hypersensitivity to semaglutide
18. Other causes of hyperandrogenism (example: tumor, CAH) or amenorrhea (untreated thyroid disease, tumor, primary ovarian failure, prolactinoma).
19. Active symptoms or undergoing treatment for anorexia nervosa or binging/purging disorder

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Cree-Green, MD, PhD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- University of Colorado Anshutz Medical Campus/Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 5 participants who screen failed, and 4 participants who withdrew due to not tolerating the study medication.
Period: Overall Study
Arm/Group | Diet Intervention | GLP-1 Intervention
Started | 17 | 43
Completed | 17 | 34
Not Completed | 0 | 9
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Screen Failure | 0 | 5

BASELINE CHARACTERISTICS:
Population: 12-21 year old participabnts with polycystic ovary syndrome
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet Intervention | GLP-1 Intervention | Total
Number analyzed (Participants) | 17 | 38 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.44 (1.55) | 15.65 (1.71) | 15.20 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 38 | 55
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 18 | 27
  Not Hispanic or Latino | 8 | 20 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 38 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Fat Fraction
Description: Change from baseline in presence/severity of hepatic fat fraction will be measured with MRI, and calculated via the Dixon method as the proton density hepatic fat fraction, which ranges from 0-75%. A negative value means a decrease in liver fat, and a positive value means an increase in liver fat.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Change in percentage of liver fat
Arm/Group | Diet Intervention | GLP-1 Intervention
Number analyzed (Participants) | 17 | 34
Change in percentage of liver fat | -1.41 (2.24) | -1.84 (4.39)

2. Primary Outcome: Change in Weight
Description: Change in weight will be calculated for each group (diet and semaglutide), and both the absolute and relative weight changes between the two groups will be reported.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Change in weight (KG)
Arm/Group | Diet Intervention | GLP-1 Intervention
Number analyzed (Participants) | 17 | 34
Change in weight (KG) | -1.66 (2.81) | -5.30 (4.92)

3. Secondary Outcome: Change in Rate of De Novo Lipogenesis (DNL)
Description: Change from baseline of the rate of overnight de novo lipogenesis (DNL) will be measured utilizing stable isotope methods with deuterated water, and expressed as the rate of newly synthesized lipids in the serum triglyceride fraction. A negative value means a decrease in newly synthesized lipids after the 12 week intervention, and a positive value means an increase in newly synthesized lipids after the 12 week intervention. A lower value is better.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Diet Intervention | GLP-1 Intervention
Number analyzed (Participants) | 17 | 34
mg/dL | 0.94 (5.7) | -1.9 (1.0)

4. Secondary Outcome: Change in Whole Body Insulin Sensitivity
Description: Participants will undergo a 75 gram oral glucose tolerance test, and the change from baseline in whole body insulin sensitivity will be expressed as Si, calculated via the oral minimal model.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: dl/kg/min per microU/ml
Arm/Group | Diet Intervention | GLP-1 Intervention
Number analyzed (Participants) | 17 | 34
dl/kg/min per microU/ml | 0.0000629 (0.000193) | 0.000213 (0.000423)

5. Secondary Outcome: Change in Adipose Insulin Sensitivity
Description: Change from baseline of adipose insulin sensitivity will be calculated as the percent suppression of free fatty acids, and the nadir of free fatty acids during the oral glucose tolerance test. Percent suppression of FFAs during the OGTT was calculated as fasting FFA minus the minimal FFA value divided by fasting FFA. This was calculated for baseline and after 12-weeks of intervention. The change was calculated by subtracting the final-baseline values. A higher absolute value means there was an improvement in adipose insulin sensitivity after 12-weeks of treatment.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Diet Intervention | GLP-1 Intervention
Number analyzed (Participants) | 17 | 34
percentage of change | 0.44 (12.06) | -1.431 (9.97)

6. Other Pre Specified Outcome: Change in Percentage of Indirect Glycerol Carbon Contributions to Newly Synthesized Triglycerides and Glucose
Description: This outcome evaluates mitochondrial function and excess tricarboxylic acid (TCA) cycle substrate cycling by measuring indirect carbon contributions to newly synthesized triglycerides and glucose using stable isotope-labeled glycerol. Participants receive orally administered [U-13C3]glycerol mixed in water, and plasma glucose and lipids are analyzed by 13C NMR spectroscopy. Indirect glycerol carbon contribution reflects the fraction of glycerol carbons that first enter the TCA cycle before incorporation into triglycerides and glucose. A decrease in the percentage of indirect contributions is beneficial, indicating decreased oxidative stress resulting from excess TCA cycling.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of indirect glycerol carbon c
Arm/Group | Diet Intervention | GLP-1 Intervention
Number analyzed (Participants) | 17 | 34
percentage of indirect glycerol carbon c | -1.59 (3.19) | 3.08 (5.24)

7. Other Pre Specified Outcome: Change in Free Androgen Index
Description: The Free Androgen Index (FAI) is a test for hyperandrogenism in women, using testosterone and sex hormone binding globulin (SHBG) as markers. The calculation is FAI = Total Testosterone (nmol/ L)) x 100 / Sex Hormone-Binding Globulin (SHBG) (nmol/ L). Typical values for the FAI in women are 7-10, and FAI is usually elevated in women with PCOS. The change in FAI will be calculated after 12 weeks of diet or semaglutide intervention. A negative value means an improvement as there was a decrease in androgen levels after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Diet Intervention | GLP-1 Intervention
Number analyzed (Participants) | 17 | 34
unitless | -3.05 (4.94) | -2.45 (3.27)

ADVERSE EVENTS:
Time Frame: Measured up to 4 months from enrollment
Arm/Group | Diet Intervention | GLP-1 Intervention
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/38
Other Adverse Events (participants affected / at risk) | 0/17 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT03919929/Prot_SAP_000.pdf